CLINICAL TRIAL: NCT06345404
Title: A Phase 1, Randomized, Blinded, Placebo-controlled, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, and Preliminary Efficacy of ITK Inhibitor Soquelitinib in Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Safety, Tolerability, and Preliminary Efficacy of Soquelitinib in Participants With Moderate to Severe AD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-818-003
Record Dates: First submitted 2024-03-12; First posted 2024-04-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Sequential Dose Escalation and Dose Expansion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Soquelitinib Dose Escalation and Dose Expansion (Experimental): In Dose Escalation, participants will receive soquelitinib tablets orally at one of three dose levels (100 mg twice daily, 200 mg once daily, 200 mg twice daily) for 28 days.
  In Dose Expansion, participants will receive soquelitinib tablets orally at a dose selected from the dose escalation part of the study, for 56 days
  Interventions: Drug: Soquelitinib
- Placebo (Placebo Comparator): Participants in the Dose Escalation part of the study will receive placebo tablets orally once daily or twice daily for 28 days.
  Participants in the Dose Expansion part of the study will receive placebo tablets orally once daily or twice daily for 56 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Soquelitinib — Tablets
  Arms: Soquelitinib Dose Escalation and Dose Expansion
Drug: Placebo — Soquelitinib matching placebo tablets
  Arms: Placebo

SUMMARY:
Safety, tolerability, and preliminary efficacy of soquelitinib in participants with moderate to severe AD

DETAILED DESCRIPTION:
A Phase 1, Randomized, Blinded, Placebo-controlled, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, and Preliminary Efficacy of ITK Inhibitor Soquelitinib in Participants with Moderate to Severe Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, ≥18 years of age at Screening.
2. Atopic dermatitis, according to Hanifin and Rajka criteria and confirmed by a dermatologist.
3. Moderate to severe disease defined by EASI ≥16; body surface area ≥10; and vIGA ≥3.
4. Documented history of inadequate response or intolerance to one or more topical therapies (including but not limited to corticosteroids, immune modulators, PDE-4 inhibitors) and/or systemic therapies (including but not limited to, dupilumab, cyclosporine, mycophenolate, azathioprine, oral corticosteroids or a JAK inhibitor, e.g., tofacitinib, baricitinib, and ruxolitinib).
5. A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period.
6. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after last dose of study treatment

Exclusion Criteria:

1. Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis, cutaneous lupus, previous burns, or extensive tattoos) that would interfere with evaluations of the effect of study medication on AD.
2. Other active skin diseases or skin infections (bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline visit or would interfere with the appropriate assessment of AD lesions.
3. Administration of oral prednisone or its equivalent within 2 weeks of starting the trial or receiving corticosteroids parenterally within 4 weeks of Screening.
4. Administration of oral or injectable immunosuppressive medications such as methotrexate, mycophenolate, azathioprine, cyclosporine, dupixent, a janus kinase inhibitor or tacrolimus (except that topical is allowed) within 4 weeks of Screening.
5. Active use of phototherapy, attending a tanning booth, or extended sun exposure which could affect judging disease activity.
6. Female participant who is pregnant, breastfeeding or is considering becoming pregnant during the study or for approximately 120 days after the last dose of study intervention.
7. Male participant who is considering fathering a child or donating sperm during the study or for approximately 120 days after the last dose of study intervention.
8. History of immunosuppression not related to medication (such as common variable hypogammaglobulinemia), history of clinically significant medical conditions (such as anemia, neutropenia, thrombocytopenia, abnormal renal function, or abnormal liver function), planned surgical procedures, or any other reason which in the opinion of the investigator or Sponsor would interfere with the participant's participation in this study, would make the participant an unsuitable candidate to receive study intervention, or would put the participant at risk by participating in the protocol; or permanently wheelchair-bound or bedridden or very poor functional status which prevents the ability to perform self-care.
9. Have an unstable or uncontrolled illness, including but not limited to cerebrocardiovascular (e.g., unstable angina, unstable arterial hypertension, moderate to severe heart failure [New York Heart Association Class III/IV]), respiratory, gastrointestinal, endocrine, hematologic, or neurologic disorders that would potentially affect participant safety within the study or confound efficacy and safety assessments.
10. Participants with renal function which is moderately or severely impaired, defined as an estimated glomerular filtration rate (eGFR) ≤59 ml/minute.
11. Participants with abnormal liver function as recognized by the FDA and as defined by the Child-Pugh criteria. Specifically, participants must show no signs of encephalopathy, have no ascites, have a serum bilirubin ≤2.0 mg/dL, have a serum albumin ≥3.5 g/dL, and have a prothrombin time prolonged by no more than 4 seconds.
12. Any of the following laboratory values would preclude participation in this trial:

    * Hematocrit <30%
    * Neutrophil count <2000/μl
    * Liver enzymes ≥2 × upper limit of normal (ULN)
    * Platelet count <100,000/μl
13. Participants who cannot ingest medications orally or who have malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, changes in laboratory values, vital signs, and electrocardiograms | Up to 30 days after last intervention administration
  Incidence, nature, and severity of treatment-emergent adverse events of soquelitinib compared with placebo, including changes in laboratory values, vital signs, and electrocardiograms (ECGs)

SECONDARY OUTCOMES:
To determine the efficacy of soquelitinib in participants with atopic dermatitis as measured by percent change in Eczema and Severity Index (EASI) | Up to 90 days after last intervention administration
  The Eczema Area and Severity Index (EASI) is used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
To determine the efficacy of soquelitinib in participants with atopic dermatitis as measured by change in percent reaching validated Investigator Global Assessment (vIGA) of 0 or 1 | Up to 90 days after last intervention administration
  The vIGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema, induration/papulation, lichenification and oozing/crusting, and takes extent of disease into account. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Mahabhashyam, MD, Study Director — Corvus Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Clinical Site 5, Birmingham, Alabama
  - Clinical Site 9, Tucson, Arizona
  - Clinical Site 3, North Little Rock, Arkansas
  - Clinical Site 2, Fremont, California
  - Clinical Site 7, Palo Alto, California
  - Clinical Site 13, Pomona, California
  - Clinical Site 10, Castle Rock, Colorado
  - Clinical Site 6, Tampa, Florida
  - Clinical Site 11, Brooklyn, New York
  - Clinical Site 16, New York, New York
  - Clinical Site 12, New York, New York
  - Clinical Site 15, Mayfield Heights, Ohio
  - Clinical Site 1, Camp Hill, Pennsylvania
  - Clinical Site 8, Philadelphia, Pennsylvania
  - Clinical Site 4, Frisco, Texas
  - Clinical Site 14, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No